CLINICAL TRIAL: NCT02610348
Title: Persistence of Anti-Hep B Antibodies at 12 to 18 Months of Age in Children Having Received Hep B Vaccine at Birth and a DTaP-IPV-HB-Hib Hexavalent Vaccine (Hexaxim® or Infanrix Hexa®) Concomitantly With Prevnar® at 2, 4 and 6 Months of Age
Brief Title: Anti-Hep B Antibodies at Age 12 to 18 Months After Hep B Vaccine at Birth and DTaP-IPV-Hep B-PRP-T Hexavalent Vaccine Concomitantly With Prevnar® at 2, 4 and 6 Months of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A3L47; U1111-1161-2649 (Other: WHO)
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Hexaxim®; Hexyon®; Hexacima®; Prevnar®; DTaP-IPV-HB-Hib hexavalent vaccine
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Toddlers vaccinated with Hexaxim®/Hexyon®/Hexacima® in study A3L12
  Interventions: Biological: DTaP-IPV-HB-PRP~T and Pneumococcal polysaccharide vaccines
- Group B (Experimental): Toddlers vaccinated with Infanrix hexa® in study A3L12
  Interventions: Biological: DTaP-HB-IPV and Pneumococcal polysaccharide vaccines

INTERVENTIONS:
Biological: DTaP-IPV-HB-PRP~T and Pneumococcal polysaccharide vaccines — Original Vaccine in Study A3L12 (NCT00401531). No vaccination will be administered as part of this study
  Arms: Group A
Biological: DTaP-HB-IPV and Pneumococcal polysaccharide vaccines — Original Vaccine in Study A3L12 (NCT00401531). No vaccination will be administered as part of this study
  Arms: Group B

SUMMARY:
Primary Objective:

To describe the persistence of Hep B antibodies (Ab) at 12 to 18 months of age following a three-dose infant primary series vaccination of either Hexaxim®/Hexyon®/Hexacima® or Infanrix® hexa at 2, 4 and 6 months of age following Hep B vaccination at birth.

DETAILED DESCRIPTION:
Sera from subjects who have participated in study PNA19 trial (NCT00594347) and for whom parents or legal representatives had given authorization to use the sera taken from their child will be used for this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having received 4 Hep B doses in A3L12 (i.e. one dose at birth + three doses during study at 2, 4 & 6 months of age)
* Subjects having participated in PNA19
* Subject's parents having given authorization to use serum collected in PNA19 for future research
* The initials, birth date, and gender of the subject are consistent between A3L12 and PNA19 databases
* Subjects for whom retention sera are of enough volume to allow a valid determination of the HBsAg antibody level.

Exclusion Criteria:

* Not applicable.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Levels of anti-Hepatitis B antibody concentrations in subject that received Hexaxim® or Infanrix® hexa vaccine in a previous study | Day 0
  Levels of anti-Hepatitis B antibody concentrations will be determined at ≥ 10 mIU/mL and ≥ 100 mIU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (2):
- Thailand (2):
  - Bangkok
  - Khon Kaen

REFERENCES:
- [Result] Kosalaraksa P, Chokephaibulkit K, Benjaponpitak S, Pancharoen C, Chuenkitmongkol S, B'Chir S, Da Costa X, Vidor E. Persistence of hepatitis B immune memory until 9-10 years of age following hepatitis B vaccination at birth and DTaP-IPV-HB-PRP approximately T vaccination at 2, 4 and 6 months. Hum Vaccin Immunother. 2018 May 4;14(5):1257-1265. doi: 10.1080/21645515.2018.1426418. Epub 2018 Feb 21. PMID 29333947